CLINICAL TRIAL: NCT00428311
Title: The Cardiovascular Risk Profile Associated With The Polycystic Ovary Syndrome And With Ovulatory Hyperandrogenism, And Its Changes During Treatment With Metformin Or Oral Contraceptives
Brief Title: Effects of Metformin vs Oral Contraceptives on CV Risk Markers in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOPCOS 01/2003
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-31 (Estimated); Status verified 2007-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Hyperandrogenism; Hirsutism; Cardiovascular risk; Chronic inflammation; Metformin; Cyproterone acetate; Oral contraceptives
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Hirsutism | interventions — Metformin; Ethinyl Estradiol; Cyproterone Acetate

INTERVENTIONS:
Drug: Metformin
Drug: Ethynyl-estradiol plus cyproterone acetate

SUMMARY:
Cardiovascular risk factors cluster in hyperandrogenic women - including those presenting with the polycystic ovary syndrome - in association with insulin resistance, obesity, and other metabolic disorders.

The present clinical trial intends to compare the effects of oral contraceptives and metformin on PCOS patients, focusing on classic and non-classic cardiovascular risk markers and indexes of cardiovascular performance, in order to whether or not, as suspected by previous data obtained in non-hyperandrogenic women, oral contraceptives worsen the cardiovascular risk profile of PCOS women, favoring the use of metformin if the latter actually ameliorates such a risk.

ELIGIBILITY:
Inclusion Criteria:

* Women of fertile age presenting with PCOS
* Non-hyperandrogenic women of fertile age (these women will not receive the interventions and will serve only to obtain normative data for some variables)

Exclusion Criteria:

* Severe disease not related to the condition under study
* Pregnancy
* Medical or surgical treatment of PCOS during the previous 3 months
* Contraindication for the use of oral contraceptives or metformin
* Inability to understand the proposal of the study precluding effective informed consent
* Minors who are not accompanied by their legal representative

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2004-04; Study Completion 2006-10

PRIMARY OUTCOMES:
Serum androgen levels
Lipid profiles
Blood pressure
Cardiovascular performance
Non-classic cardiovascular risk markers
Indexes of insulin secretion and sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Héctor F Escobar-Morreale, MD, PhD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Department of Endocrinology, Hospital Ramón y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Luque-Ramirez M, Escobar-Morreale HF. Treatment of polycystic ovary syndrome (PCOS) with metformin ameliorates insulin resistance in parallel with the decrease of serum interleukin-6 concentrations. Horm Metab Res. 2010 Oct;42(11):815-20. doi: 10.1055/s-0030-1262855. Epub 2010 Aug 20. PMID 20730705
- [Derived] Luque-Ramirez M, Alvarez-Blasco F, Escobar-Morreale HF. Antiandrogenic contraceptives increase serum adiponectin in obese polycystic ovary syndrome patients. Obesity (Silver Spring). 2009 Jan;17(1):3-9. doi: 10.1038/oby.2008.491. Epub 2008 Nov 6. PMID 18997670
- [Derived] Luque-Ramirez M, Alvarez-Blasco F, Uriol Rivera MG, Escobar-Morreale HF. Serum uric acid concentration as non-classic cardiovascular risk factor in women with polycystic ovary syndrome: effect of treatment with ethinyl-estradiol plus cyproterone acetate versus metformin. Hum Reprod. 2008 Jul;23(7):1594-601. doi: 10.1093/humrep/den095. Epub 2008 Mar 27. PMID 18375410
- [Derived] Luque-Ramirez M, Alvarez-Blasco F, Botella-Carretero JI, Sanchon R, San Millan JL, Escobar-Morreale HF. Increased body iron stores of obese women with polycystic ovary syndrome are a consequence of insulin resistance and hyperinsulinism and are not a result of reduced menstrual losses. Diabetes Care. 2007 Sep;30(9):2309-13. doi: 10.2337/dc07-0642. Epub 2007 May 29. PMID 17536071